CLINICAL TRIAL: NCT06296069
Title: Cognitive-motor Training on a Labile Surface in Stroke Inpatients: Feasibility and Preliminary Effects
Brief Title: Exergames on an Unstable Surface in Stroke Inpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eleftheria Giannouli (Other)
Responsible Party: Sponsor-Investigator, Eleftheria Giannouli, Dr., Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SwingIT-stroke
Record Dates: First submitted 2024-02-20; First posted 2024-03-06 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Stroke
Keywords: exergames; cognitive-motor; proprioception; stroke; motor-cognitive; inpatient rehabilitation; neurologic patients; cognition; balance; gait; technology-based training; exercise; serious games; active video games
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The intervention group will conduct an exergame-based cognitive-motor intervention on a unstable surface (on top of their standard inpatient treatment).
  Intervention duration will be tailored to the stay in the inpatient rehabilitation clinic (3-4 weeks). Training sessions will last 20-28 minutes (progressive increase).
  Interventions: Other: exergame-based cognitive-motor training on an unstable surface
- Control group (Active Comparator): The intervention group will conduct an exergame-based cognitive-motor intervention on a stable surface (on top of their standard inpatient treatment).
  Intervention duration will be tailored to the stay in the inpatient rehabilitation clinic (3-4 weeks). Training sessions will last 20-28 minutes (progressive increase).
  Interventions: Other: exergame-based cognitive-motor training on an stable surface

INTERVENTIONS:
Other: exergame-based cognitive-motor training on an unstable surface — The intervention group will receive an exergame-based cognitive-sensorimotor intervention on an unstable surface (by placing the exergame device (Senso) on an unstable surface).
  The Senso is a platform for the dynamic recording of steps, weight shifts and other body movements producing forces. For the labile condition, the Senso is mounted on steel balls, allowing the platform to swing freely along the horizontal plane. There is no movement induced by the platform itself. Sway is only induced when the participant steps and shifts the center of pressure. The degree of instability and movement of the platform can be adjusted by inducing a dampening. The dampening can be set manually, either to on or off. When damping is on, the movement can be reduced by predefined percentages. The maximum displacement of the platform is thereby 100 mm to each side.
  Arms: Intervention group
Other: exergame-based cognitive-motor training on an stable surface — The control group will receive an exergame-based cognitive-motor intervention on an stable surface using the exergame device Senso.
  The Senso is a platform for the dynamic recording of steps, weight shifts and other body movements producing forces.
  Arms: Control group

SUMMARY:
Aim of this study is to assess the feasibility and effects of exergame-based cognitive-motor training on a labile platform on physical and cognitive functioning in stroke inpatients.

This is two-armed pilot randomized controlled trial taking place in an inpatient neurologic rehabilitation clinic. A total of 30 persons that are undergoing inpatient rehabilitation due to a stroke will be randomly assigned to either the intervention group (IG) or the control group (CG). Participants of the IG will receive exergame-based motor-cognitive training on a labile surface, whereas participants of the CG will train on a stable surface. Primary outcome is feasibility comprising measures of adherence, attrition, safety and usability. Secondary outcomes will be measures of cognitive (psychomotor speed, inhibition, selective attention, cognitive flexibility, brain activity) and motor (functional mobility, gait speed, balance, proprioception) functioning.

DETAILED DESCRIPTION:
As a result of the impairment in cognitive and motor functioning after a stroke, the balance ability worsens and gait becomes unsteady. Of all complications following a stroke, falls are one of the most prevalent and the frequency of total fall events is rising with time after the stroke. Since falls are in general the leading reason for injuries in older adults and about a third of persons older than 65 years fall once a year, there is an overall need for interventions.

Balance training is an established form of exercise in people suffering from stroke and other neurological disabilities. However, cognitive-motor training is superior to single physical training in improving motor functioning e.g. gait speed and walking endurance in stroke patients. More specifically, compared to sequential (e.g. cycling followed by cognitive training) and simultaneous-additional (e.g. cycling while solving an arithmetical task), simultaneous-incorporated motor-cognitive training (e.g. any type of training in which the cognitive task is "incorporated" into the motor task, i.e. the cognitive task is a relevant prerequisite to successfully solve the motor-cognitive task) seems to be the most promising training type for improving gait speed and potentially other functions in stroke patients.

Exergames (interactive (cognitive) games which are played by body movements) are an excellent tool for the delivery of simultaneous-incorporated cognitive-motor training and they have already been used in the context of several frail and neurologic populations, including stroke patients.

Proprioception is used to stabilize the body by sensing its position in space via the sense of joint and limb positioning. Proprioception training addresses the balance and somatosensory stimulation and can therefore build a possible prevention strategy for further falls and of managing ADLs. Combining proprioceptive training with simultaneous cognitive tasks could have additional positive outcomes in stroke rehabilitation. Indeed, a recent systematic review concluded that proprioceptive and dual-task exercises stimulate and promote postural balance, gait, and quality of life and reduce the risk of falls in stroke patients compared with traditional rehabilitation programs.

There is currently just one study that has looked into the effects of exergame-based cognitive-motor training with the additional proprioceptive stimulation (by playing the exergames on a labile platform). They found that compared to the training on a stable platform and to a passive control group, training on an instable platform is more effective for the improvement of reactive balance and functional mobility under dual-task conditions in healthy, community-dwelling older adults. The feasibility and effects of this type of training (exergame training on labile surface and thus rich in proprioceptive stimulation) in stroke patients remains unknown.

Therefore, the aim of this study is to assess the feasibility and effects of exergame-based cognitive-motor training on a labile platform on physical and cognitive functioning in stroke inpatients.

The investigators hypothesize that exergame-based cognitive-motor on a labile surface will be feasible within the context of inpatient rehabilitation of stroke patients. In addition, the investigators hypothesize that compared to training on stable surface, training on a labile platform will be more effective for the improvement of motor and cognitive functioning in stroke inpatients.

This is two-armed pilot randomized controlled trial taking place in an inpatient neurologic rehabilitation clinic. A total of 30 persons that are undergoing inpatient rehabilitation due to a stroke will be randomly assigned to either the intervention group (IG) or the control group (CG). Participants of the IG will receive exergame-based motor-cognitive training on a labile surface, whereas participants of the CG will train on a stable surface. Primary outcome is feasibility comprising measures of adherence, attrition, safety and usability. Secondary outcomes will be measures of cognitive (psychomotor speed, inhibition, selective attention, cognitive flexibility, brain activity) and motor (functional mobility, gait speed, balance, proprioception) functioning.

ELIGIBILITY:
Inclusion Criteria:

* Prescription for inpatient rehabilitation due to a stroke
* Ability to provide a signed informed consent
* Mini-Mental State Examination (MMSE) score ≥ 20
* Physically able to stand for at least 3 minutes without external support (self-report)

Exclusion Criteria:

* Insufficient knowledge of the German language to understand the instructions and the games
* Conservatively treated osteoporotic fractures in the last 16 weeks
* Depending on assistance for ambulation (Functional Ambulation Categories <2),
* Mobility, cognitive, sensory and/or psychiatric limitations or comorbidities which impair the ability to play the exergames and/or conduct the pre-/post assessments

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2024-09-17 (Actual)

PRIMARY OUTCOMES:
Security incidents | through study completion, an average of 6 months (over all training sessions)]
  Total number of (Serious) Adverse Events (SAE/AE)
Attrition rate | through study completion, an average of 6 months
  Number of Drop-outs as percentages of patients included in the study
Adherence rate | through study completion, an average of 6 months (over all training sessions)]
  Number of attended training sessions as percentages of total possible training sessions
Usability | The System Usability Scale is recorded at the end of the training period and as part of the T2 measurements, through study completion (max. 6 months)
  Usability will be assessed on basis of the validated German version of the System Usability Scale (SUS-DE). The SUS-DE is assessed in week 6 of the exergame-based intervention. It consists of ten items that are rated on a five-point Likert scale (i.e. ranging from 1 - "strongly disagree" to 5 - "strongly agree"). A total score will be calculated according to the scoring guidelines of the SUS. The total SUS score ranges between 0 and 100, whereas higher scores indicate better usability. A total SUS score of at least 70 will be considered an "acceptable" solution (i.e. 52 = ok, 73 = good, 85 = excellent, 100 = best imaginable).
Training Load | The 2 questions of the Nasa-TLX will be asked after each training session, through study completion (about 6 months). Answers will be presented descriptively for each training session as well as aggregated by averaging values across all training sessions
  The NASA-Task Load Index (TLX) is a self-report, multidimensional assessment tool that rates perceived workload in order to assess a task, a system, or other aspects of performance (in this case the exergames). It contains five subscales: Mental Demand, Physical Demand, Temporal Demand, Performance, Effort and Frustration. Each subscale can be given a score between 0 and 20. A higher score reflects a higher workload. For this study only the 2 subscales "Mental Demand" and "Physical Demand" will be used.
Enjoyment | The EEQ is recorded at the end of the training period and as part of the T2 measurements, through study completion (about 6 months)
  Enjoyment of the exergame-based intervention concept will be assessed on basis of the Exergame Enjoyment Questionnaire (EEQ) that will be translated to German according to the guidelines for the process of cross-cultural adaptation of self-report measures. It consists of 20 statements corresponding to four categories of questions: (1) immersion, (2) intrinsically rewarding activity, (3) control, and (4) exercise. Each statement will be responded to on a five-point Likert scale (i.e. strongly disagree (1 point), disagree (2 points), neutral (3 points), agree (4 points), and strongly agree (5 points). The EEQ will be analyzed by calculating the average overall score as well as an average score for each category of questions.
User experience | The User Experience questions is recorded at the end of the training period and as part of the T2 measurements, through study completion (about 6 months)
  Several questions specifically tailored to this study regarding perceived safety, perceived positive effects, intention to recommend etc. will be used. Most questions will have a 7step Likert Scale answers. However, there will also be two open ended questions asking for any positive/negative feedback and other general remarks by the participants.
Training Goals | The GAS will be defined at T1 (baseline) and will be reevaluated in the middle (after 8 trainings) and T2 (post assessments), through study completion (about 6 months)
  Personal goals regarding rehabilitation/training will be assessed with the Goal Attainment Scale (GAS). The GAS is an individual approach to defining and evaluating personal rehabilitation goals. The scale consists of a five-point rating of the achievement of the specified goals. A score of 0 corresponds to the expected improvement or achievement of the predefined goal. A negative score of -1 or -2 is considered worse than expected. A positive score of 1 and 2 is given when the goal is achieved even better than expected. Interpersonal scores for the three time-points will be evaluated descriptively for each participant separately.

SECONDARY OUTCOMES:
Changes in cognitive flexibility | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within 2 days prior to starting or after completing the intervention
  Cognitive flexibility will be assessed using the Trail making test (TMT): The TMT is a widely used neuropsychological test only requiring paper and pencil and has two parts, TMT.A and TMT.B. Circled numbers from 1 to 25 are allocated randomly on a sheet which participants have to connect in the right order (TMT.A). At TMT-B, circled numbers and letters are randomly allocated on a sheet and the participants have to connect circled numbers and letters in the right order and in alternating manner. The required time to complete each task as well as the difference between the scores TMT.B-TMT.A measured in both parts will be evaluated.
Changes in psychomotor speed | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within 2 days prior to starting or after completing the intervention
  The Step Reaction Time Test measures psychomotor speed in terms of reaction to visual stimuli using the lower extremities in 6 directions (front right, front left, right, left, back right & back left). There are six light grey triangles on the screen and each time one of then turns black, participants need to step as quickly as possible in the respective direction. Average reaction time across all stimuli will be used for analyses.
Changes in selective attention | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within 2 days prior to starting or after completing the intervention
  The Go/No-Go test measures selective attention and inhibition. Participants fixate on a small grey dot in the middle of the screen. Crosses (+) and Xs (x) appear on the right and left side of the grey dot in a randomised order. The task is to ignore the + and just conduct a step as quickly as possible in the direction that an (x) appears.
Changes in inhibition and brain activity | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within 2 days prior to starting or after completing the intervention
  The Stroop Test assesses inhibition. A computer-based version of the Stroop Colour-Word will be conducted. Participants are instructed to press a button corresponding to the ink or colour of the ink/color of the word/stimuli that appears on the screen as quickly as possible. Reaction time in ms on response-correct trials and accuracy in % is extracted separately for compatible and incompatible trials. The Stroop Test will be coupled with functional a near-infrared spectroscopy (fNIRS) system (NIRx Medical Technologies, NIRSport2, Berlin, Germany) to assess which brain regions are active during the cognitive test. Outcomes are the average change from baseline concentration of Oxyhaemoglobin (HbO2) and haemoglobin (HHb) with no cognitive task in comparison to conducting a cognitive test (Stroop). Another outcome builds the difference from the peak concentration of HbO2 to the baseline with no cognitive task.
Changes in functional mobility | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within 2 days prior to starting or after completing the intervention
  Functional mobility will be measured using the instrumented version of the Timed Up and Go Test (iTUG). Four inertial sensor units (Opal, APDM, Oregon USA) are attached to the participant's body. At the start signal participants must stand up from a chair, walk 3 meters at a comfortable walking speed, come back and sit down on the chair again. A dual-task condition will also be conducted. In the dual-task condition participants have to count backwards in steps of three from a random given number while they are performing the test. Following outcome measures will be used for further analyses for the single task and the dual-task conditions respectively: total duration, sit-to-stand duration, turn velocity, turn-to-sit velocity. Additionally, relative dual task costs (DTC) of walking as percentage of loss relative to the single-task walking performance, according to the formula DTC [%] = 100 * (single-task score - dual-task score)/single-task score will be calculated.
Changes in coordination | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within 2 days prior to starting or after completing the intervention
  Motor coordination is assessed using the 4 Step Square test (4SST). The 4SST assess a person's ability to step as quickly as possible in all 4 directions: forward, backward and sidewards. At the start, the participant stands in Square 1, facing Square 2 and will step clockwise over every Square until Square 4 and anti- clockwise back to Square 1. Time is measured to complete this task.
Changes in dynamic balance | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within 2 days prior to starting or after completing the intervention
  Dynamic balance is assessed with the Shape Tracking Test. Participants are asked to move their center of pressure (COP) displacement by bending or rotating their body without moving the feet, so that they remain within the track that is shown on the screen.
Changes in static balance | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within 2 days prior to starting or after completing the intervention
  Postural Sway will be assessed with the iSway test of the APDM inertial sensor system. One inertial sensor unit (Opal, APDM, Oregon USA) is attached to the participant's body (lower back) with an elastic strap. Participants are required to stand as still as possible for 30 seconds. Several center of pressure (COP) displacement measures are computed with the Software "Mobility Lab 2®; Oregon", that comes along with the inertial sensor system. Mean displacement velocity and sway area will be used for further analyses.
Changes in gait | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within 2 days prior to starting or after completing the intervention
  Gait Analysis will be conducted with the iWalk test of the APDM inertial sensor system. Four inertial sensor units (Opal, APDM, Oregon USA) (two at the feet, one at the lower back and one on the chest) are attached to the participant's body with elastic straps. Participants are required to walk for 2 minutes. Two trials will be conducted for each participant: on in their preferred walking speed and one in which participants are asked to walk as fast as possible (but without running). Several gait performances metrics are computed with the software "Mobility Lab 2®; Oregon, that comes along with the inertial sensor system. Stride length, stride velocity, and gait variability will be used for further analyses.
Changes in leg proprioception | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within 2 days prior to starting or after completing the intervention
  Leg proprioception will be assessed using the ProMeTo-System. In this test, the examiner will move participants joints into several positions. Participants will be asked to memorize and replicate exactly the position that the examiner specified without visual control. Average angle differences for each joint will be used for further analyses.
  Because there are currently no reference values and/or standard error measurement values for this population, this test will be repeated twice before the onset of the intervention (once during the pre-assessment, together with all the rest of the pre-port assessments and once again one day later, just before starting the first training session) in order to calculate its test-retest reliability and assessment error (minimum detectable difference) for this population.
Changes in balance confidence | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within 2 days prior to starting or after completing the intervention
  The German version of the Activity- specific balance confidence scale (ABC-D) will be used to assess balance confidence in various activities in older people. The questionnaire uses a scale from 0 to 100% about the confidence of maintaining balance by activities. In total sixteen questions will be asked, and the total mean scores will be calculated.
Changes in gait confidence | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within 2 days prior to starting or after completing the intervention
  The German version of the Modified gait efficacy scale (mGES-D) will be used to assess perception of confidence in walking under challenging circumstances. It is a 10-item questionnaire on a 10- point Likert scale. 1 means no confidence; 10 means full confidence. 100 points means complete confidence in every task.

CONTACTS AND LOCATIONS:
Overall Officials: Eleftheria Giannouli, PhD, Principal Investigator — ETH Zurich
Locations (1):
- Rehaklinik Zihlschlacht, Zihlschlacht-Sitterdorf, Thurgau, Switzerland

REFERENCES:
- [Background] Abbott RD, Curb JD, Rodriguez BL, Masaki KH, Popper JS, Ross GW, Petrovitch H. Age-related changes in risk factor effects on the incidence of thromboembolic and hemorrhagic stroke. J Clin Epidemiol. 2003 May;56(5):479-86. doi: 10.1016/s0895-4356(02)00611-x. PMID 12812823
- [Background] Katan M, Luft A. Global Burden of Stroke. Semin Neurol. 2018 Apr;38(2):208-211. doi: 10.1055/s-0038-1649503. Epub 2018 May 23. PMID 29791947
- [Background] Chen X, Liu F, Lin S, Yu L, Lin R. Effects of Virtual Reality Rehabilitation Training on Cognitive Function and Activities of Daily Living of Patients With Poststroke Cognitive Impairment: A Systematic Review and Meta-Analysis. Arch Phys Med Rehabil. 2022 Jul;103(7):1422-1435. doi: 10.1016/j.apmr.2022.03.012. Epub 2022 Apr 10. PMID 35417757
- [Background] Lipardo DS, Tsang WWN. Falls prevention through physical and cognitive training (falls PACT) in older adults with mild cognitive impairment: a randomized controlled trial protocol. BMC Geriatr. 2018 Aug 24;18(1):193. doi: 10.1186/s12877-018-0868-2. PMID 30143002
- [Background] Chiaramonte R, Bonfiglio M, Leonforte P, Coltraro GL, Guerrera CS, Vecchio M. Proprioceptive and Dual-Task Training: The Key of Stroke Rehabilitation, A Systematic Review. J Funct Morphol Kinesiol. 2022 Jul 7;7(3):53. doi: 10.3390/jfmk7030053. PMID 35893327
- [Background] Mura G, Carta MG, Sancassiani F, Machado S, Prosperini L. Active exergames to improve cognitive functioning in neurological disabilities: a systematic review and meta-analysis. Eur J Phys Rehabil Med. 2018 Jun;54(3):450-462. doi: 10.23736/S1973-9087.17.04680-9. Epub 2017 Oct 25. PMID 29072042
- [Background] Wuest S, van de Langenberg R, de Bruin ED. Design considerations for a theory-driven exergame-based rehabilitation program to improve walking of persons with stroke. Eur Rev Aging Phys Act. 2014;11(2):119-129. doi: 10.1007/s11556-013-0136-6. Epub 2013 Dec 7. PMID 25309631
- [Background] Jaggi S, Wachter A, Adcock M, de Bruin ED, Moller JC, Marks D, Schweinfurther R, Giannouli E. Feasibility and effects of cognitive-motor exergames on fall risk factors in typical and atypical Parkinson's inpatients: a randomized controlled pilot study. Eur J Med Res. 2023 Jan 16;28(1):30. doi: 10.1186/s40001-022-00963-x. PMID 36647177
- [Background] Altorfer P, Adcock M, de Bruin ED, Graf F, Giannouli E. Feasibility of Cognitive-Motor Exergames in Geriatric Inpatient Rehabilitation: A Pilot Randomized Controlled Study. Front Aging Neurosci. 2021 Nov 29;13:739948. doi: 10.3389/fnagi.2021.739948. eCollection 2021. PMID 34912206
- [Background] Subramaniam S, Wang S, Bhatt T. Dance-based exergaming on postural stability and kinematics in people with chronic stroke - A preliminary study. Physiother Theory Pract. 2022 Nov;38(13):2714-2726. doi: 10.1080/09593985.2021.1994072. Epub 2021 Dec 2. PMID 34852719
- [Background] Morat M, Bakker J, Hammes V, Morat T, Giannouli E, Zijlstra W, Donath L. Effects of stepping exergames under stable versus unstable conditions on balance and strength in healthy community-dwelling older adults: A three-armed randomized controlled trial. Exp Gerontol. 2019 Nov;127:110719. doi: 10.1016/j.exger.2019.110719. Epub 2019 Sep 9. PMID 31513877
- [Background] Brooke, J., SUS: A quick and dirty usability scale. Usability Eval. Ind., 1995. 189.
- [Background] Lohmann, K. and J. Schäffer, System Usability Scale (SUS)-An Improved German Translation of the Questionnaire, 2013. URL https://minds. coremedia. com/2013/09/18/sus-scale-an-improved-german-translation-questionnaire, 2015.
- [Background] Bangor, A., P. Kortum, and J. Miller, Determining What Individual SUS Scores Mean: Adding an Adjective Rating Scale. J. Usability Stud., 2009. 4: p. 114-123.
- [Background] Hart, S., Nasa-task load index (Nasa-TLX); 20 years later. Vol. 50. 2006.
- [Background] Bowie CR, Harvey PD. Administration and interpretation of the Trail Making Test. Nat Protoc. 2006;1(5):2277-81. doi: 10.1038/nprot.2006.390. PMID 17406468
- [Background] Reitan, R.M., Validity of the Trail Making Test as an Indicator of Organic Brain Damage. Perceptual and Motor Skills, 1958. 8(3): p. 271-276.
- [Background] Tombaugh TN. Trail Making Test A and B: normative data stratified by age and education. Arch Clin Neuropsychol. 2004 Mar;19(2):203-14. doi: 10.1016/S0887-6177(03)00039-8. PMID 15010086
- [Background] Zimmermann, P. and B. Fimm, A test battery for attentional performance. Applied neuropsychology of attention. Theory, diagnosis and rehabilitation, 2002. 110: p. 151.
- [Background] Salarian A, Horak FB, Zampieri C, Carlson-Kuhta P, Nutt JG, Aminian K. iTUG, a sensitive and reliable measure of mobility. IEEE Trans Neural Syst Rehabil Eng. 2010 Jun;18(3):303-10. doi: 10.1109/TNSRE.2010.2047606. Epub 2010 Apr 12. PMID 20388604
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Wright DL, Kemp TL. The dual-task methodology and assessing the attentional demands of ambulation with walking devices. Phys Ther. 1992 Apr;72(4):306-12; discussion 313-5. doi: 10.1093/ptj/72.4.306. PMID 1584862
- [Background] Wulf G, McNevin N, Shea CH. The automaticity of complex motor skill learning as a function of attentional focus. Q J Exp Psychol A. 2001 Nov;54(4):1143-54. doi: 10.1080/713756012. PMID 11765737
- [Background] Mancini M, King L, Salarian A, Holmstrom L, McNames J, Horak FB. Mobility Lab to Assess Balance and Gait with Synchronized Body-worn Sensors. J Bioeng Biomed Sci. 2011 Dec 12;Suppl 1:007. doi: 10.4172/2155-9538.S1-007. PMID 24955286
- [Background] Mancini M, Salarian A, Carlson-Kuhta P, Zampieri C, King L, Chiari L, Horak FB. ISway: a sensitive, valid and reliable measure of postural control. J Neuroeng Rehabil. 2012 Aug 22;9:59. doi: 10.1186/1743-0003-9-59. PMID 22913719
- [Background] Dite W, Temple VA. A clinical test of stepping and change of direction to identify multiple falling older adults. Arch Phys Med Rehabil. 2002 Nov;83(11):1566-71. doi: 10.1053/apmr.2002.35469. PMID 12422327
- [Background] Schott N. [German adaptation of the "Activities-Specific Balance Confidence (ABC) scale" for the assessment of falls-related self-efficacy]. Z Gerontol Geriatr. 2008 Dec;41(6):475-85. doi: 10.1007/s00391-007-0504-9. German. PMID 18327692
- [Background] Altmeier D, Giannouli E. German translation and psychometric properties of the modified Gait Efficacy Scale (mGES). Z Gerontol Geriatr. 2020 May;53(3):251-255. doi: 10.1007/s00391-019-01507-5. Epub 2019 Feb 6. PMID 30725165
- [Background] Scarpina F, Tagini S. The Stroop Color and Word Test. Front Psychol. 2017 Apr 12;8:557. doi: 10.3389/fpsyg.2017.00557. eCollection 2017. PMID 28446889
- [Derived] Buttiker J, Marks D, Hanke M, Ludyga S, Marsico P, Eggimann B, Giannouli E. Cognitive-motor exergame training on a labile surface in stroke inpatients: study protocol for a randomized controlled trial. Front Neurol. 2024 Jun 19;15:1402145. doi: 10.3389/fneur.2024.1402145. eCollection 2024. PMID 38966081